CLINICAL TRIAL: NCT07173569
Title: St Mary's Assisted Reproductive Technology and Cardiometabolic Health: Modifiable Targets for Multimorbidity Prevention (START-HEALThY)
Acronym: START-HEALThY
Status: Not yet recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Lucy Higgins, Senior Clinical Lecturer and Honorary Consultant Obstetrician, University of Manchester
Other Study IDs: 351318
Record Dates: First submitted 2025-07-14; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Maternal Cardiometabolic Health; Infertility; Assisted Reproductive Technology; Cardiovascular Health; Metabolic Health; in Vitro Fertilisation
Keywords: Feasibility study; Ambulatory cardiometabolic health monitoring; Cohort
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood serum samples, with participant consent, will be retained for the length of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-conception: history of infertility cohort: Individuals with a history of infertility who have been accepted to undergo in vitro fertiliitsation (IVF) treatment (NHS or private funding) at the Department of Reproductive Medicine, Manchester University NHS Foundation Trust.
- Pre- conception: no history of infertility cohort: Healthy individuals with no history of infertility, attending a pre-conception appointment at Manchester University NHS Foundation Trust.
- Post-pregnancy cohort: Individuals who participated in the START (St Mary's After Reproductive Technology) clinic study (20/NE/0220) who consented to receive future research invitations, will be invited to a research appointment 1-5 years post-birth.

SUMMARY:
The main causes of death in women are conditions affecting the heart and blood vessels (cardiovascular disease, CVD). Women who have difficulties getting pregnant (infertility) may be at increased risk, but the reasons for this are not clear. Infertility itself may be linked with poorer heart and blood vessel health, or fertility treatments such as in vitro fertilisation (IVF) could increase the risk.

The study aims to understand the practicalities of obtaining detailed profiling of women's pre- and post- pregnancy heart, blood vessel and metabolic health. Two groups of women in Manchester University NHS Foundation Trust, will be recruited over 2 years: 1) women planning a pregnancy, either spontaneously or with IVF treatment after infertility, 2) women who previously took part in a pregnancy health study after IVF or non-IVF conception.

Participants will attend a single research appointment where they will undergo a cardiometabolic health assessment. They will have their BMI calculated, body composition measured, a measurement of how well their blood vessels work using a blood pressure cuff around the arm and/or finger and blood sampling performed. A blood pressure cuff as well as a blood sugar sensor may be fitted to be worn after the appointment. Participants will be asked to complete a questionnaire(s), with follow-up for up to 13 months.

The cardiometabolic health of those who conceived with or without IVF treatment and with or without a history of infertility will be compared at both time points to investigate the possibility of links between infertility, IVF processes and CVD risk and to understand any potential barriers to recruitment of individuals at either time point to guide future studies. This information could then be used in a full-scale study, including in pregnancy, to improve care and promote lifelong health for women with infertility.

DETAILED DESCRIPTION:
Objectives:

Primary objective: To assess the feasibility of a pre-conception and postnatal cardiometabolic health research study in infertile and fertile individuals.

Secondary objectives:

* To assess clinic-measured cardiometabolic status
* To measure ambulatory cardiovascular status
* To measure ambulatory blood glucose concentrations
* To assess the views of fertile and infertile individuals on cardiometabolic health optimisation and research in this area
* To assess acceptability of cardiometabolic status measurement approaches (clinic and ambulatory measured) in fertile and infertile populations
* To conduct initial exploratory investigations into whether cardiometabolic status is influenced by a history of infertility

Study Design This is a prospective observational cohort study consisting of two cohorts: a pre-conception cohort and a post-pregnancy cohort made up of individuals with and without a history of infertility. All participants of either cohort will have one research visit.

Individuals will be invited to attend a single face-to-face research appointment where the following will be undertaken:

* • Electronic wwritten consent will be obtained by a GCP-trained member of the clinical research team and a study number allocated.
* Optional consent will be obtained for access to medical records held at MFT (pertaining to any subsequent pregnancy and cardiometabolic outcomes, if in the pre-conception cohort) and to future data linkage studies related to future cardiometabolic health outcomes.
* Demographic data, medical history including cardiovascular/metabolic/obstetric/gynaecological history, medication history as well as mental health history, diet, breastfeeding, exercise, education and smoking status will be recorded.
* Anthropometric measurements, including height, weight, lean and fat mass (bioimpedance scale) and adiposity distribution (skin fold thickness), will be measured. BMI and waist-hip ratio will be calculated.
* Non-invasive assessments of cardiovascular function will be performed, including Mobil-O-Graph (pulse wave velocity, cardiac output, blood pressure, heart rate and total vascular resistance) using a blood pressure cuff, with or without EndoPAT 2000™ (endothelial function and vascular stiffness) via finger probes before and after occlusion with a blood pressure cuff.
* Blood samples (maximum 15ml of blood, equivalent to six teaspoons) for assessment of renal function, lipid levels and glucose control via HbA1C, will be collected by an appropriately trained member of the research team, analysed and clinically reported in line with routine clinical care.
* An ambulatory blood pressure monitor/pulse wave analyser (Mobil-O-Graph) will be fitted (if consent provided and a machine is available) and participants requested to wear this for 24 hours following the appointment, while conducting their daily activities. Once the Mobil-O-Graph device is returned the data will be downloaded by a member of the clinical research team and analysed.
* A continuous glucose monitor (CGM; FreeStyle Libre Pro IQ) will be fitted (if consent provided and a machine is available) and participants requested to wear for a minimum of 24-48 hours following the appointment, while conducting their daily activities (CGM data can be collected from a single sensor for up to 14 days). CGM data will be downloaded once the device is returned.

Participants will be asked to complete a post-participation questionnaire during the visit or via an email link sent to the participant after the visit, exploring:

* Views on cardiometabolic health optimisation
* Acceptability of the cardiometabolic health assessment, timing, approach to investigation and overall acceptability of participation

Analysis:

As this is a feasibility study, analysis will be through descriptive statistics (e.g., means/medians, standard deviations/interquartile ranges for continuous variables and frequencies and percentages for categorical variables) precision estimates (i.e., width of confidence interval).

We will conduct exploratory regression analyses to inform the design of adequately powered future studies.

Potential impact:

This study will assess the feasibility of recruiting individuals, with/without an infertility history, to a study of pre-conception and postnatal cardiometabolic status assessment. It will give initial indications of whether any difference in cardiometabolic health of infertile individuals pre-dates IVF treatment and/or persists or resolves in the short-term post-delivery. It will be the first to use ambulatory measures of cardiometabolic health (such as wearable blood pressure and glucose monitors), which may have increased sensitivity to detect subtle signs of (differences in) cardiometabolic (dys)function during normal activity, compared with single time point measures during clinical visits.

Ultimately, a better understanding of cardiometabolic dysfunction in infertile individuals may enable pre- or post- conception intervention (dietary, exercise and potentially pharmacological treatment) to optimise health before, during and after pregnancy in a life course approach to women's health (with anticipated positive impacts on the health of any resulting infant(s)).

ELIGIBILITY:
Inclusion Criteria:

* In pre-conception cohort:

  * Aged between 16 and 45
  * Able to provide informed consent
  * Either: 1) Those with a history of infertility (failure to conceive after at least 1 year of unprotected intercourse/3-6 cycles of Intra-Uterine Insemination (IUI) or diagnosed cause of infertility) and accepted for IVF at The Department of Reproductive Medicine, MFT or, 2) attending for a pre-conception appointment at MFT
  * Nulliparous (no previous pregnancies beyond 20 weeks)
  * No pre-existing heart disease, hypertensive disease, vascular disease or diabetes
* In post-pregnancy cohort

  * Aged between 16 and 45
  * Able to provide informed consent
  * Participant of START clinic study (achieved pregnancy via a) IVF with or without ICSI treatment, b) spontaneous conception without medical intervention within 12 months, or c) spontaneous conception following ovulation induction for delay in spontaneous conception >12 months or confirmed anovulation)

Exclusion Criteria:

- In all participants:

* Prisoners
* Born male at birth
* Language barrier not overcome by telephone or video interpretation services
* Pregnant at time of study visit

Pre-conception participants only:

• Accepted for IVF for non-infertility reasons i.e. egg donation, egg collection, egg banking, gestational surrogacy

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: There are two cohorts for this study: pre-conception and post-pregnancy.
  For the pre-conception cohort of the study, two groups of participants will be recruited:
  * Group 1: individuals with a history of infertility who have been accepted to undergo IVF treatment at the Department of Reproductive Medicine, MFT.
  * Group 2: individuals with no history of infertility, attending for a pre-conception appointment at MFT.
  For the post-pregnancy cohort of the study, individuals who participated in the START (St Mary's After Reproductive Technology) clinic study (20/NE/0220) who consented to receive future research invitations, will be invited to an research appointment at 1-5 years post-birth.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment | Through study duration, approximately 23 months
  Number of recruits

SECONDARY OUTCOMES:
Recruitment acceptance | Through study duration, approximately 23 months
  Proportion of eligible individuals accepting recruitment
Time taken to achieve the proposed sample size | Recruitment period, approximately 23 months
  Time taken to achieve the proposed sample size
Acceptance of the investigative methods | Through study duration, approximately 23 months
  Proportion of individuals accepting each type of investigation
Duration of ambulatory monitoring | Up to 14 days post-study visit
  Duration of ambulatory monitoring completed per participant
Consent to data linkage | Through study duration, approximately 23 months
  Proportion of individuals consenting to data linkage
Participant questionnaire asking about importance of cardiometabolic health optimisation and research in this area | Through study duration, approximately 23 months
  Participant-reported importance of cardiometabolic health optimisation and research in this area via electronic questionnaire. Participants will be asked to rank on a Likert scale (strongly disagree to strongly agree) whether they would consider taking part in a similar study in the future, whether they would recommend the study to a friend, whether the research topic is important to them and would they improve their health if they knew their cardiometabolic health was below average.
Participant questionnaire asking about acceptability of participation and of measurement techniques in the study | Through study duration, approximately 23 months
  Participant-reported acceptability of participation and of individual measurements. Participants will be asked to rank on a Likert scale (strongly disagree to strongly agree) how they felt about the acceptability of measurements performed in clinic as well as ambulatory measurements (if applicable).
Variability between cohort differences in cardiometabolic health markers | Following analysis of data, an average of 3 years from study start
  Preliminary variability between cohort differences in cardiometabolic health markers, to identify potential useful investigations for future studies. Example health markers include adiposity differences (BMI, waist-hip ratio), non-invasive assessments of cardiovascular function (in-clinic and ambulatory Mobil-O-Graph results), serum renal function, lipid levels and HbA1C and ambulatory CGM measurements.
Proportion of pre-conception participants who conceive within a year of the study visit | A year after participant's study visit
  Proportion of pre-conception participants who conceive within a year of the study visit